CLINICAL TRIAL: NCT06694025
Title: Post-marketing Surveillance Study for the Safety of Efluelda Tetra Pre-filled Syringe, a High-dose Quadrivalent Influenza Vaccine Administered to Adults 65 Years or Older in the Republic of Korea.
Brief Title: Post-marketing Surveillance Study for the Safety of Efluelda Tetra Pre-filled Syringe.
Status: Not yet recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: QHD00024; U1111-1251-6083 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Immunization; Influenza (Healthy Volunteers)
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Efluelda group: A single dose of 0.7 mL is administered as approved by MFDS.
  Interventions: Biological: Efluelda Tetra Pre-filled syringe

INTERVENTIONS:
Biological: Efluelda Tetra Pre-filled syringe — Suspension for injection in a pre-filled syringe

SUMMARY:
To investigate the incidence of adverse events (AEs) and adverse drug reactions (ADRs) occurred following administration of Efluelda Tetra in adults aged 65 years or older under routine clinical practice, as per approved indications.

The study duration of each participation will be approximately 28 to 35 days. In the event that Visit 2 is not made, the study duration would be extended to 36 to 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years or older on the day of enrollment
* The informed consent form has been signed and dated
* Receipt of 1 dose of Efluelda Tetra on the day of enrollment according to the approved local product label

Exclusion Criteria:

* Previous history of enrollment in this study
* Participation at the time of study enrollment (or in the 4 weeks preceding the enrollment) or planned participation during the present study period in a clinical study investigating a vaccine, drug, medical device or medical procedure

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Investigators will recruit participants after vaccination with Efluelda Tetra as per routine healthcare visits and according to approved local product labeling, at study centers (general hospitals or clinics located in Korea).
Sampling Method: Non-Probability Sample
Enrollment: 670 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of solicited (pre-listed in the participant's diary card [DC] and case report form) injection site and systemic reactions | From baseline up to 7 days after vaccination
Occurrence of unsolicited AEs and ADRs | From baseline up to Visit 2 (28-35 days) after vaccination
Occurrence of unexpected AEs and ADRs | From baseline up to participant's last contact after vaccination (36-42 days)
Occurrence of serious adverse events (SAEs) and serious adverse drug reactions (SADRs) | From baseline up to participant's last contact after vaccination (36-42 days)
Occurrence of AE of special interest (AESI) | From baseline up to participant's last contact after vaccination (36-42 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number : 001, Seoul, Seoul-teukbyeolsi, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org